CLINICAL TRIAL: NCT06944652
Title: Flexibility Training (Stretching) to Improve Jumping Performance
Brief Title: Stretching to Improve Jumping Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4925
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Vertical Jump Performance

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are being masked as to the study hypothesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plantar flexor stretching (Experimental): Flexibility training (stretching) of the muscles at the back of the lower leg
  Interventions: Other: Stretching
- Shoulder stretching (Active Comparator): Flexibility training (stretching) of the muscles surrounding the shoulder joint
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Stretching — Stretching of the plantar flexors or the shoulder joint

SUMMARY:
The study involves comparison of an 8-week plantar flexor stretching program to a shoulder stretching program for improving vertical jump performance in adolescent athletes.

DETAILED DESCRIPTION:
Increasing flexibility may improve vertical jump performance. For example, being able to go deeper into a squat before jumping may allow for greater force development through the range of movement and this may transfer to greater vertical jump height. The study compares plantar flexor stretching to shoulder stretching for improving vertical jump performance in adolescent athletes. Athletes are being stratified by sex and maturity status (before or after estimated age at peak height velocity) and randomized to one of two groups: Plantar flexor stretching (2 sets of 6 stretches, 5 times per week) or the same volume of shoulder stretching. Before and after training, participants are being assessed for vertical jump and landing performance.

ELIGIBILITY:
Inclusion Criteria:

* Currently involved in a sport training program

Exclusion Criteria:

* Current or past injuries that might affect jumping performance or stretching the plantar flexors or shoulder joint

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Counter movement jump height | Change over 8 weeks
  Counter movement jump height assessed on a force plate

SECONDARY OUTCOMES:
Take-off velocity | Change over 8 weeks
  Take-off velocity assessed on a force plate in the right and left limbs
Ground reaction force on take off | Change over 8 weeks
  Ground reaction force on take off from a counter movement jump on a force plate in right and left limbs
Ground reaction force on landing | Change over 8 weeks
  Ground reaction force when landing from a jumping on force plate in right and left limbs
Ground reaction force when landing from a standard height | Change over 8 weeks
  Ground reaction force when landing from a height (150% of baseline counter movement jump height)
Functional dorsiflexor range of movement | Change over 8 weeks
  Functional dorsiflexor range of movement assessed with an inclinometer in left and right limbs
Active dorsiflexor range of movement | Change over 8 weeks
  Active dorsiflexor range of movement assessed with a goniometer in right and left limbs
Passive dorsiflexor range of movement | Change over 8 weeks
  Passive dorsiflexor range of movement assessed with a goniometer in right and left limbs
Shoulder flexibility | Change over 8 weeks
  Shoulder flexibility assessed with a goniometer in right and left limbs

CONTACTS AND LOCATIONS:
Locations (1):
- College of Kinesiology University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No